CLINICAL TRIAL: NCT02638285
Title: Pregnancy Rate by HCG Administration Versus Urinary LH Surge Method in Patients Undergoing IUI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Payam Peymani, Head Of Pharmacoepidemiology Department, Health policy Research Center,Shiraz university of Medical Sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShirazSUMSnew
Record Dates: First submitted 2015-12-16; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Pregnancy
MeSH Terms: interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HCG group (Experimental): HCG group
  Interventions: Drug: HCG; Drug: Clomiphene
- LH group (Experimental): LH group
  Interventions: Drug: LH; Drug: Clomiphene
- clomiphene citrate (Experimental): clomiphene citrate
  Interventions: Drug: LH; Drug: HCG

INTERVENTIONS:
Drug: LH
  Arms: LH group; clomiphene citrate
Drug: HCG
  Arms: HCG group; clomiphene citrate
Drug: Clomiphene
  Arms: HCG group; LH group

SUMMARY:
To compare pregnancy rate by Human Chorionic Gonadotropin (HCG) administration and urinary Luteinizing Hormone (LH) surge method for insemination in patients undergoing Intrauterine Insemination (IUI) at Montaserieh infertility center.

The present study comprised 309 infertile women candidate for IUI, randomly divided into LH surge and HCG groups (assign the number for each patient, odds number for LH and even number for HCG group). All patients were subjected to baseline ultrasound and received clomiphene citrate before undergoing serial transvaginal sonography. LH was measured using LH kit when 2-5 follicles (18-20 mm) appeared in LH surge group, and if positive, IUI was performed after 24 hours. In HCG group, the patients received HCG 1000 units and underwent IUI after 36 hours. The pregnancy rate was then compared in LH and HCG groups.

ELIGIBILITY:
Inclusion Criteria:

* infertile women candidate for IUI

Exclusion Criteria:

* women with negative urinary LH surge which required HCG administration,
* those with more than 5 follicles who had to use LH kit and not receive HCG to avoid ovarian hyperstimulation.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | Two weeks after IUI

CONTACTS AND LOCATIONS:
Locations (1):
- Health Policy Research Center, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Yes